CLINICAL TRIAL: NCT03910855
Title: Investigating the Impact of Mindfulness on Psychological Well-being of Stroke Survivors and Their Caregivers: A Randomized Controlled Trial.
Brief Title: Impact of Mindfulness on Psychological Well-being of Stroke Survivors and Their Caregivers
Acronym: SOMII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201711-00071
Record Dates: First submitted 2019-02-12; First posted 2019-04-10 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Stress; Anxiety; Depression
Keywords: Mindfulness; Stroke Survivors; Caregivers
MeSH Terms: conditions — Stroke; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either a Mindfulness-based Intervention (MBI) or a Health Education Program (HEP). The intervention is for 4 weeks. Measures will be administered prior to and on completion of the intervention, and at 3-month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Intervention (Experimental): The mindfulness-based intervention consists of four 2-hour sessions covering various mindfulness techniques (e.g. mindfulness of breath, body and movement, senses and informal practice, and empathy and compassion) that pertain to stroke survivors and their family caregivers. Participants will be provided handouts for the information covered during these talks and discussions.
  Interventions: Behavioral: Mindfulness Based Intervention
- Health Education Program (Active Comparator): The health education program consists of four 2-hour sessions covering various health topics (e.g. diet, nutrition and exercise) that pertain to stroke survivors. Participants will be provided handouts for the information covered during these talks and discussions.
  Interventions: Other: Health Education Program

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — The mindfulness-based intervention consists of four 2-hour sessions covering various mindfulness techniques (e.g. mindfulness of breath, body and movement, senses and informal practice, and empathy and compassion) that pertain to stroke survivors and their family caregivers. Participants will be provided handouts for the information covered during these talks and discussions.
  Arms: Mindfulness Based Intervention
Other: Health Education Program — The health education program consists of four 2-hour sessions covering various health topics (e.g. diet, nutrition and exercise) that pertain to stroke survivors. Participants will be provided handouts for the information covered during these talks and discussions.
  Arms: Health Education Program

SUMMARY:
This study will employ a randomized control design. Stroke survivors and family caregivers will be recruited for the study, and randomized either to receive mindfulness-based intervention or health education. Both programs consist of 4 2-hour sessions. Participants of the mindfulness-based intervention (MBI) will be taught and guided in practice of psychosocial interventions that are focused on (1) stress management and coping skills, (2), body awareness and movement, (3) feelings of empathy and compassion and (4) motivation for rehabilitation. Participants of the health education program (HEP) will learn and discuss topics related to self-care and post-stroke management. Measures will be administered prior to and on completion of the intervention, and at 3-month follow-up. They will be used to assess symptoms associated with depression, anxiety, stress, perceived quality of life and participant characteristics such as personality variables.

DETAILED DESCRIPTION:
Stroke prevalence is 3-4% among Singaporeans above the age of 50, and will rise with our aging population. Stroke survivors face many concerns, including physical, psychological, cognitive and psychosocial consequences of stroke, as well as impaired functioning and quality of life. They often rely on their family for physical, cognitive and emotional support in order to perform daily functional activities. Dependence on family members has been shown to affect the physical, mental and emotional well-being of caregivers of stroke survivors. Research indicates that the long-term demands of caring for a stroke survivor puts a strain on caregivers who may not be able to provide the appropriate amount of care required to manage the needs of stroke survivors over time.

Mindfulness-based interventions (MBIs) are increasingly being offered as psychotherapeutic interventions for individuals who suffer from medical conditions such as stroke, and for their long-term family caregivers. Several review studies have shown that MBIs, specifically for long-term conditions, enhanced the ability to cope with physical difficulties, improved mental and emotional well-being as well as overall quality of life, promoting better health outcomes. A systematic review investigating the use of MBIs with stroke survivors found that psychological, physiological and psychosocial outcomes were improved, such as anxiety, depression, mental fatigue and overall quality of life (Lawrence et al., 2013).

However, there are limited data for stroke survivors and their caregivers especially among Asians. Furthermore, there is little attention to study the interaction between participants characteristics and MBIs to determine whether there are any specific moderators that help to maximize the therapeutic outcomes of MBIs (Shaprio et al., 2011). Although there are growing number of studies correlating personality traits and dispositional mindfulness (Hanley, 2016; Giluk, 2009), little research has been done to examine personality traits as moderators to treatment outcome. Research focusing the the five-factor model of personality has demonstrated that the five personality traits have different strengths of correlation with the dispositional mindfulness. Among the traits, neuroticism displayed the strongest negative correlation with depositional mindfulness while conscientiousness displayed the strongest positive correlation with depositional mindfulness.

This study will be the first to examine the moderating effects of personality traits on the impact of mindfulness-based intervention in terms of depression, anxiety, stress and perceived quality of life of stroke survivors and their family caregivers. Furthermore, this study will evaluate and compare the impacts of mindfulness-based intervention and health education on the psychological well-being of both the participants. Findings will encourage the development of future strategies to understand the variability in treatment response and prognosis as well as to address individual differences with relevant psychotherapy skills.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors and/ or their
* Family Caregivers
* Comprehends and provides consent independently

Exclusion Criteria:

-Cognitively impaired individuals with a MMSE score of less than 20, and a MoCA score of less than 23.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Cohen Perceived Stress Scale, PSS | An average of 1 Month
  A 10-item measure evaluating the perception of stress.
Centre for Epidemiologic Studies Depression Scale (CES-D) | An average of 1 Week
  A 20-item measure for epidemiological research on depression.
Stroke Specific Quality of Life Scale (SS-QOL) | An average of 1 month
  A 49-item self-report questionnaire designed to measure the heath related quality of life specific to stroke survivors across 12 domains.
Stroke Impact Scale (SIS) | An average of 1 week
  A 64-item questionnaire that assesses across 8 domains
Short-Form-36 (SF-36) | A range from 4 to 52 weeks
  A 36-item self-report survey of health, including physical and mental health. Higher scaled scores reflect better quality of health.
The State-Trait Anxiety Inventory, STAI | State: Current state, Trait: An average of 1 month
  The STAI is a commonly used measure of trait and state anxiety.

SECONDARY OUTCOMES:
Zarit Burden Inventory (ZBI) | An average of 1 month
  A 22-item self-report questionnaire to measure for level of caregiver burden or stress.
The Big Five Personality Inventory, BFI | An average of 1 month
  44-item inventory that measures an individual on the Big Five Factors (dimensions) of personality.
Five Facet Mindfulness Questionnaire, FFMQ | An average of 1 month
  This 39-item instrument is based on a factor analytic study of five independently developed mindfulness questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Kinjal Doshi, PhD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Preliminary data to inform design of future studies.